CLINICAL TRIAL: NCT04195412
Title: Neuroplasticity Following Bihemispheric Transcranial Direct Current Stimulation and Motor Training in Chronic Stroke Patients.
Brief Title: Imaging the Effects of Bihemispheric Transcranial Stimulation and Motor Training After Stroke.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRJ1913
Record Dates: First submitted 2019-10-29; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: Stroke Rehabilitation; Transcranial Direct Current Stimulation; Neuroimaging; Neuronal Plasticity
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (Experimental): Bihemispheric tDCS will be applied. The anode will be placed on the affected hemisphere, while the cathode will be positioned over the unaffected hemisphere. After stimulation, individual and intensive upper limb rehabilitation will be performed.
  Interventions: Device: tDCS + upper limb rehabilitation
- Control (Sham Comparator): Bihemispheric sham tDCS will be applied. The anode will be placed on the affected hemisphere, while the cathode will be positioned over the unaffected hemisphere. After sham stimulation, individual and intensive upper limb rehabilitation will be performed.
  Interventions: Device: Sham tDCS + upper limb rehabilitation

INTERVENTIONS:
Device: tDCS + upper limb rehabilitation — Stimulation will be applied for 20 minutes by a DC stimulator (NeuroConn, Germany). During each stimulation section, a pair of saline-soaked sponge electrodes (surface 24 cm²) will be placed over C3 and C4, according to the International 10-20 EEG system. Stimulation intensity will be 2 mA with current ramping up and down of 10 seconds each. The stimulation will be followed by 40 minutes of upper limb rehabilitation. Experimental sessions will be repeated five times per week to complete 10 sessions.
  Arms: tDCS
Device: Sham tDCS + upper limb rehabilitation — Sham stimulation will be applied for 20 minutes by a DC stimulator (NeuroConn, Germany). During each sham stimulation section, a pair of saline-soaked sponge electrodes (surface 24 cm²) will be placed over C3 and C4, according to the International 10-20 EEG system. The anode will be placed to the affected hemisphere, while the cathode will be positioned over the unaffected hemisphere. Sham tDCS will be performed by ramping current flow for the first 10 seconds of stimulation, but switching the stimulator off automatically after 30 seconds. The sham stimulation will be followed by 40 minutes of upper limb rehabilitation. Experimental sessions will be repeated five times per week to complete 10 sessions.
  Arms: Control

SUMMARY:
Functional and structural magnetic resonance imaging (MRI) will be used to investigate neural correlates of bihemispheric transcranial direct current stimulation (tDCS) associated with upper limb rehabilitation in chronic stroke patients. For this purpose, patients included will be submitted to 10 sessions with active or sham bihemispheric tDCS associated with intensive and individualized rehabilitation. Neuroimage will be employed before and after the intervention to investigate neural correlates of expected changes in motor function.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Stroke (> 12 months)
* Upper limb sensorimotor sequelae due to stroke affecting only one cerebral hemisphere
* The structural integrity of the corpus callosum sensorimotor
* Showing ability to perform some movement with the paretic upper limb: at least minimal active mobility of the wrist and two fingers of the paretic hand.
* Score ≥ 18 at Folstein Mini-Mental State Examination

Exclusion Criteria:

* Score ≥ 4 at Ashworth Scale
* MRI or tDCS contraindications (cardiac pacemakers; implanted medication pumps; cochlear, or eye implants; craniotomy, skin lesions at the site of stimulation; surgical clips in or near the brain; claustrophobia, history of seizures, permanent makeup or tattoos with metallic dyes…)
* Prior neurological diseases
* Hemodynamic instability
* Pregnancy
* Traumatic or orthopedic lesion limiting the range of upper limb motion
* Severe comprehension deficits, apraxia or neglect that would interfere with performing the study tasks
* Score > 59 at the Fugl-Meyer Assessment of Motor Recovery after Stroke

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Treatment-related changes in functional magnetic resonance imaging | pre-treatment (baseline), post-treatment (from 3 to 7 days after the end of the treatment)
  Brain functional changes from baseline to post-treatment
Treatment-related changes in white matter | pre-treatment (baseline), post-treatment (from 3 to 7 days after the end of the treatment)
  Brain structural (white matter) changes from baseline to post-treatment

SECONDARY OUTCOMES:
Changes in Fugl-Meyer assessment of paretic upper limb motor function | pre-treatment (baseline), post-treatment (from 3 to 7 days after the end of the treatment); 30 days follow up (30 days after completing treatment) and 90 days follow up (90 days after completing treatment)
  Fugl-Meyer Upper Extremity (FM-UE) Scale of Motor Impairment scores changes from baseline to post-treatment, 30 and 90 days later (follow up).
Changes in Jebsen-Taylor Hand Function Test scores | pre-treatment (baseline), post-treatment (from 3 to 7 days after the end of the treatment), follow-up 30 days, follow-up 90 days
  Fugl-Meyer Upper Extremity (FM-UE) Scale of Motor Impairment scores changes from baseline to post-treatment and in subsequent follow-up
Changes in Stroke Impact Scale scores | pre-treatment (baseline), post-treatment (from 3 to 7 days after the end of the treatment), follow-up 30 days, follow-up 90 days
  Stroke Impact Scale scores changes from baseline to post-treatment and in subsequent follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda F Tovar-Moll, PhD, Study Director — D'Or Institute for Research and Education (IDOR); Erika C Rodrigues, PhD, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- D'Or Institute for Research and Education (IDOR), Rio de Janeiro, Brazil